CLINICAL TRIAL: NCT06116812
Title: The Effects of Laughter Yoga and Mindfulness-based Stress Reduction (MBSR) Practices Applied to Women With Breast Cancer Receiving Chemotherapy on Anxiety, Depression, Quality of Life and Spiritual Well-being Levels: A Randomized Controlled Study
Brief Title: The Effects of Laughter Yoga and Mindfulness-Based Stress Reduction (MBSR) Practices Applied to Women With Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafkas University (Other)
Responsible Party: Principal Investigator, Zehra Coktay, PhD Student, Kafkas University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 04578878
Record Dates: First submitted 2023-10-31; First posted 2023-11-03 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer; Laughter Therapy; Mindfulness Therapy; Life Quality; Anxiety and Depression; Spiritual Well-being
MeSH Terms: conditions — Breast Neoplasms; Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- the laughter yoga group (Experimental): Women diagnosed with breast cancer who meet the inclusion criteria and are receiving chemotherapy will receive laughter therapy twice a week for an average of 40-60 minutes for 8 weeks.
  Interventions: Other: the laughter yoga group
- the mindfulness based stress reduction group (Experimental): Women diagnosed with breast cancer who meet the inclusion criteria and are receiving chemotherapy will receive an average of 40-60 minutes of mindfulnes therapy twice a week for 8 weeks.
  Interventions: Other: the mindfulness based stress reduction group
- the control group (No Intervention): Women diagnosed with breast cancer who meet the inclusion criteria and are receiving chemotherapy will receive standard hospital care only.

INTERVENTIONS:
Other: the laughter yoga group — They will gather in five-person chemotherapy rooms, and laughter therapy will be applied to the women in the application group while they are receiving chemotherapy. Sessions will last approximately 40-60 minutes.The application will last for a total of 8 weeks, twice a week.
  The 9th and 16th sessions will be held face to face and the scales will be filled in face to face meetings in these weeks (at the end of the 4th week and the 8th week). Since patients receive chemotherapy treatment once a month, face-to-face sessions are planned to be administered while the patient is receiving treatment. (Those whose treatment timing frequency is not appropriate will be excluded).
  * Other sessions will be held online via smartphone applications. Online sessions will be determined according to the mutual decision of the participants, at a time convenient for the participants.
  * In the 12th week, all groups will have the scales filled in again.
  Arms: the laughter yoga group
Other: the mindfulness based stress reduction group — Mindfulnes therapy will be applied to the women in the application group while they are receiving chemotherapy, in five-person chemotherapy rooms. Sessions will last approximately 40-60 minutes.The application will last for a total of 8 weeks, twice a week.
  The 9th and 16th sessions will be held face to face and the scales will be filled in face to face meetings in these weeks (at the end of the 4th week and the 8th week). Since patients receive chemotherapy treatment once a month, face-to-face sessions are planned to be administered while the patient is receiving treatment. (Those whose treatment timing frequency is not appropriate will be excluded).
  * Other sessions will be held online via smartphone applications. Online sessions will be determined according to the mutual decision of the participants, at a time convenient for the participants.
  * In the 12th week, all groups will have the scales filled in again.
  Arms: the mindfulness based stress reduction group

SUMMARY:
Breast cancer is defined as the most common type of cancer that causes death among women (Siegel et al. 2019). It constitutes 24% of cancers and 15% of cancer-related deaths in women (T.R. Ministry of Health 2020). According to statistics made towards the end of 2020, there are 7.8 million women in the world who were diagnosed with breast cancer in the last 5 years and are alive. It is estimated that one in every 8 women will develop breast cancer in developed countries (WHO 2021).

The Ministry of Health reported the frequency of breast cancer in our country as 45.6/100,000 in women in 2018. The incidence of breast cancer is reported to be higher, especially in the 45-54 age range (TC Ministry of Health 2020).

Chemotherapy is one of the most frequently preferred treatment methods in the treatment of breast cancer and can cause serious side effects such as pain, nausea and vomiting, loss of appetite, shortness of breath, mouth sores, fatigue, insomnia, anxiety and depression, and may lead to a deterioration in the quality of life of patients (Waks and Winer 2019, Samami et al. 2021, Sajadian et al. 2017, McFarland et al. 2018, Hamer et al. 2017).

In the international and national literature, no study has been found comparing the effects of laughter and mindfulness therapy on the anxiety, depression, quality of life and spiritual well-being experienced by breast cancer patients. In this study, it is planned to investigate the effects of laughter and mindfulness therapy applications on the anxiety, depression, quality of life and spiritual well-being levels of women with breast cancer receiving chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Women who are 18 years of age or older, do not have communication problems, have and can use a smartphone, do not have internet problems to participate in group sessions, volunteer to participate in the study, receive chemotherapy at least once a month and will continue to receive chemotherapy during the study. Women with stage 1 and stage 2 breast cancer, women with primary and secondary education, women within the first year of treatment in terms of the number of cycles, women with a score of 8 or more on the Hospital anxiety and depression scale (0-7 points are normal, 8- A score of 10 is borderline, 11 and above indicates abnormality).

Exclusion Criteria:

* Women who did not meet the inclusion criteria, refused to participate in the study, and participated in less than 80% of the research practices (It is recommended to participate in at least 6 out of 8 sessions in the literature (Liu et al. 2022).),
* Women who use mindfulness therapy, laughter therapy or any complementary or integrative medicine in their daily lives outside the research, women who have a diagnosed psychological disease, metastasis or recurrence, and whose chemotherapy treatment was terminated before the study was completed,
* Women with stage 3 and stage 4 breast cancer, women who have been receiving chemotherapy for more than 1 year, women whose scores are 8 or below on the Hospital anxiety and depression scale (0-7 points indicate normal, 8-10 points indicate borderline, 11 and above indicate abnormality ).

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Since breast cancer is a type of cancer more common in women, only patients diagnosed with female breast cancer were included.
Enrollment: 105 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Hospital anxiety and depression scale outcomes | The Hospital Anxiety and Depression Scale (HADS) was developed by Zigmond and Snaith (1983). In the scale consisting of 14 items, 7 of the items measure anxiety symptoms and the other 7 measure depression symptoms.
  According to the scoring, 0-7 is considered as not sick, 8-10 is borderline sick, and 11 and above is considered seriously ill.

SECONDARY OUTCOMES:
European Organization for Research and Treatment of Cancer Quality of Life Scale (EORTC QLQ-30) outcomes | It is an assessment tool used in cancer patients and whose reliability, applicability and validity have been tested in large patient populations in 12 different countries (Björdal et al. 1999).
  Higher scores on the functional scale indicate higher/healthier functions, and higher scores on the general health status/quality of life indicate higher quality of life. However, high scores on the symptom scale indicate a high rate of symptomatology/problems (Fayers et al. 2001).
Spiritual well-being scale (Facıt-Sp-12) outcomes | The scale was developed by Peterman and his colleagues to determine the spiritual well-being of individuals with cancer and other chronic diseases (Peterman et al. 2002).
  Meaning sub-dimension (Items 2,3,5,8) has a total score of 0-16 points, Peace sub-dimension (Items 1,4,6,7) has a total score of 0-16 points, Belief sub-dimension (Items 9,10,11) ,12) total score ranges from 0-16 points, and the total score of the scale is 0-48 points. A higher scale score indicates better spiritual well-being.

CONTACTS AND LOCATIONS:
Overall Officials: zehra Coktay, phd stu, Principal Investigator — Kafkas University
Locations (1):
- Hatay Iskenderun State Hospital, İskenderun, Hatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No